CLINICAL TRIAL: NCT04212650
Title: Biologically Regulated Marrow Stimulation by Blocking Fibrosis to Improve Cartilage Repair: A Randomized Double-Blind, Placebo-Controlled Study
Brief Title: Losartan to Improve Hip Microfracture
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: redesigned trial using another placebo controlled drug
Sponsor: Steadman Philippon Research Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Office of Naval Research (ONR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-15
Record Dates: First submitted 2019-12-19; First posted 2019-12-27 (Actual); Results first posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Hip Osteoarthritis; Hip Impingement Syndrome; Cartilage Damage; Fibrosis
Keywords: Cartilage Microfracture; Losartan; Transforming growth factor beta 1; Hip Arthroscopy
MeSH Terms: conditions — Osteoarthritis, Hip; Fibrosis; Camurati-Engelmann Syndrome | interventions — Losartan

STUDY DESIGN:
Intervention Model Description: Block Randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Losartan (Experimental): 12.5mg Losartan capsules, oral administration, twice daily (25mg total per day), taken for 30 consecutive days starting on the evening of the second post-surgery day.
  Interventions: Drug: Losartan
- Placebo (Placebo Comparator): Appearance-matched placebo capsules, oral administration, twice daily, taken for 30 consecutive days starting on the evening of the second post-surgery day.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Losartan — Losartan will be administered to improve the quality of hip cartilage repair following arthroscopic microfracture. Losartan is a known anti-fibrotic agent via blocking of TGF-B1.
  Other Names: Losartan Potassium
  Arms: Losartan
Other: Placebo — Appearance-matched microcrystalline cellulose placebo
  Arms: Placebo

SUMMARY:
Phase I/IIA randomized, double-blind, placebo-controlled clinical trial to assess safety and efficacy of oral losartan for improving cartilage repair following microfracture to treat focal cartilage defects during hip arthroscopy.

DETAILED DESCRIPTION:
This is a prospective, double-blind, placebo-controlled, randomized clinical trial that will be conducted at The Steadman Clinic and Steadman Philippon Research Institute.

Articular cartilage defects that extend full thickness to subchondral bone rarely heal without intervention. Some patients may not develop clinically significant problems from acute full-thickness chondral defects, but many eventually suffer from debilitating degenerative changes. Microfracture is the most commonly used first-line treatment technique for chondral lesions in the hip, however, this procedure's effectiveness is limited by the repair tissue being a hybrid of hyaline and fibrocartilage. We hypothesize that administration of a transforming growth factor beta 1 (TGF-β1) blocker, losartan (an approved hypertension drug, angiotensin II receptor antagonist) with microfracture will enhance articular cartilage repair as assessed on quantitative magnetic resonance imaging. We will also measure patient benefit through the recording of patient reported outcomes in the 18 months following surgery. The Division of Pulmonary, Allergy and Rheumatology Products within the Center for Drug Evaluation and Research at the Food and Drug Administration has granted an investigational new drug (IND) exemption to pursue this trial in accordance with 21 CFR 312.2(b).

ELIGIBILITY:
Inclusion Criteria:

* Underwent primary hip arthroscopy
* Underwent baseline quantitative MRI at The Steadman Clinic (TSC)
* Single, localized, grade 3 or 4 cartilage lesion of the acetabulum or femoral head treated with Bone Marrow Stimulation (BMS; i.e. microfracture)
* Aged 18-60 at time of surgery
* Tonnis grade 1 or less

Exclusion Criteria:

* Two or more cartilage lesions of grade 3 or 4
* Less than 2 mm of minimal hip joint space
* Osteoarthritis or diffuse change of cartilage
* Non-English speaking
* Prior hip surgery on operative hip
* Pre-existing bony deformity caused by previous fracture(s)
* Synovial chondromatosis
* Pigmented Villonodular Synovitis (PVNS)
* Dysplasia (center edge angle <20 degrees)
* History of Avascular Necrosis (AVN), Perthes disease, or slipped capital femoral epiphysis (SCFE)
* Inflammatory arthritis or other arthritis caused by autoimmune disease
* Patients allergic to any active or inactive ingredient of losartan
* Patients taking medication with known losartan interaction, including phenobarbital, rifampin, and fluconazole.
* Subjects that are currently taking losartan

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc J Philippon, MD, Principal Investigator — Steadman Philippon Research Institute
Locations (1):
- Steadman Philippon Research Institute, Vail, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from The Steadman Clinic between March 2, 2020 and August 7, 2020. The first and last participant were enrolled on August 7, 2020.
Pre-assignment Details: Of 1 enrolled participant, 1 met inclusion criteria and was randomized to treatment.
Period: Overall Study
Arm/Group | Losartan | Placebo
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: One (1) participant was enrolled in the study and subsequently randomized to the Losartan arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan | Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: Occurrence of treatment-emergent adverse events
Time Frame: Drug related adverse events will be monitored during the medication phase (post-op days 2-31) and orthopaedic-related health and function will be monitored for the entire study duration (18 months).
Population: There was 1 subject enrolled into the Losartan arm, but withdrew before any follow-up data was collected. One serious adverse event was reported 3 days post-enrollment. This AE was determined to be unrelated to the research or study drug and is reported in the AE section.
Measure: Number; unit: participants
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 1 | 0
participants | 1 |

2. Secondary Outcome: Patient Reported Outcomes Questionnaire
Description: 12-question Short-Form General Health Survey (SF-12) - Including Physical Component Summary (PCS) and Mental Component Summary (MCS).
  * Higher score represents greater health.
  * Scale standardized to a US Population mean of 50 and standard deviation of 10 points.
Time Frame: Baseline, 3 months, 6 months, 12 months and 18 months
Population: Baseline SF-12 PCS Score was 48.8 for the 1 enrolled participant. Participant was randomized to Losartan arm but withdrew before any follow up data was collected.
Measure: Number; unit: score on a scale
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 1 | 0
score on a scale | 48.8 |

3. Secondary Outcome: Patient Reported Outcomes Questionnaire - Patient Satisfaction
Description: Patient Satisfaction
  * Scale from 1-10.
  * Higher score represents greater patient satisfaction.
Time Frame: Baseline, 3 months, 6 months, 12 months and 18 months
Population: Patient satisfaction is not collected at baseline. Participant was randomized to Losartan arm but withdrew before any follow up data was collected.
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Patient Reported Outcomes Questionnaire - Harris Hip Score
Description: Harris Hip Score (HHS).
  * Scale from 0-100.
  * Higher score represents greater hip health.
Time Frame: Baseline, 3 months, 6 months, 12 months and 18 months
Population: Baseline HHS Score was 57 for the 1 enrolled participant. Participant was randomized to Losartan arm but withdrew before any follow up data was collected.
Measure: Number; unit: score on a scale
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 1 | 0
score on a scale | 57 |

5. Secondary Outcome: Patient Reported Outcomes Questionnaire - Hip Outcome Score
Description: Hip Outcome Score (HOS) - Including Sport and Activities of Daily Living (ADL) subscales.
  * Scale from 0-100.
  * Higher score represents greater hip health.
Time Frame: Baseline, 3 months, 6 months, 12 months and 18 months
Population: Baseline HOS-ADL Score was 68 for the 1 enrolled participant. Participant was randomized to Losartan arm but withdrew before any follow up data was collected.
Measure: Number; unit: score on a scale
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 1 | 0
score on a scale | 68 |

6. Secondary Outcome: Patient Reported Outcomes Questionnaire - Western Ontario and McMaster Universities Osteoarthritis Index
Description: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) - Including Pain, Stiffness and Physical Function subscales.
  * Scale from 0-96.
  * Higher score represents worse hip health.
Time Frame: Baseline, 3 months, 6 months, 12 months and 18 months
Population: Baseline WOMAC Total Score was 31 for the 1 enrolled participant. Participant was randomized to Losartan arm but withdrew before any follow up data was collected.
Measure: Number; unit: score on a scale
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 1 | 0
score on a scale | 31 |

7. Secondary Outcome: Patient Reported Outcomes Questionnaire - Tegner Activity Scale
Description: Tegner Activity Scale
  * Scale from 0-10.
  * Higher score represents greater activity level.
Time Frame: Baseline, 3 months, 6 months, 12 months and 18 months
Population: Baseline Tegner Activity Scale was unavailable for the 1 enrolled participant. Participant was randomized to Losartan arm but withdrew before any follow up data was collected.
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Patient Reported Outcomes Questionnaire - Numeric Rating Scale for Pain
Description: Numeric Rating Scale (NRS) for Pain
  * Scale from 1-10.
  * Higher score represents greater pain.
Time Frame: Baseline, 3 months, 6 months, 12 months and 18 months
Population: Baseline NRS Pain Score was 6 for the 1 enrolled participant. Participant was randomized to Losartan arm but withdrew before any follow up data was collected.
Measure: Number; unit: score on a scale
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 1 | 0
score on a scale | 6 |

9. Secondary Outcome: Morphological and Quantitative Magnetic Resonance Imaging (MRI)
Description: Cartilage quality assessed by blinded radiologist using morphological MRI. Quantitative MRI using T2 mapping images with texture analysis used to assess water content and collagen organization within the cartilage and surrounding tissue.
Time Frame: Baseline and 12 months
Population: Participant was randomized to Losartan arm but withdrew before any follow up data was collected.
  Baseline quantitative MRI was not processed due to participant withdrawal and study closure.
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Physical Examination of the Hip - Strength
Description: Standard physical exam assessment of hip strength, measured in Newtons.
Time Frame: Baseline, 3 months, and 12 months
Population: Participant was randomized to Losartan arm but withdrew before any follow up data was collected.
  Baseline hip strength assessment data was not compiled due to participant withdrawal and study closure.
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Physical Examination of the Hip - Range of Motion
Description: Standard physical exam assessments of hip range of motion (ROM), measured in degrees.
Time Frame: Baseline, 3 months, and 12 months
Population: Participant was randomized to Losartan arm but withdrew before any follow up data was collected.
  Baseline hip range of motion assessment data was not compiled due to participant withdrawal and study closure.
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 week
Description: Participant was randomized to Losartan arm but withdrew before any follow up data was collected. Study closed.
Arm/Group | Losartan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=1) | Placebo (N=0)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient presented with increased from baseline contralateral hip pain secondary to established labral tear during a standard of care post-operative visit for the study hip, which resulted in subsequent contralateral hip surgery.

LIMITATIONS AND CAVEATS:
Per opinion of the Principal Investigator, Losartan is now clinically indicated as a standard of care post-operative therapy for patients undergoing hip microfracture surgeries. The study was terminated early, resulting in a singular subject enrolled for data analysis. The subject elected to withdraw from the study prior to the first follow-up data collection timepoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT04212650/Prot_SAP_001.pdf
  • Informed Consent Form (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT04212650/ICF_000.pdf